CLINICAL TRIAL: NCT00000798
Title: A Phase I Safety and Immunogenicity Trial of UBI Microparticulate Monovalent HIV-1 MN Peptide Immunogen in HIV-1 Seronegative Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: United Biomedical (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 018
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; Administration, Oral; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV-1 Peptide Vaccine, Microparticulate Monovalent

SUMMARY:
To evaluate the safety and immunogenicity of a new microparticulate formulation of an HIV-1 MN PND peptide for oral administration in healthy, HIV-1 seronegative adult volunteers at low risk for infection.

Vaccine formulations of synthetic peptides adsorbed to alum may not provide other requisite characteristics of an effective HIV vaccine, such as induction of mucosal immunity, production of cytotoxic T cells, and ease of administration. An oral microparticulate vaccine containing a prototype synthetic peptide has been developed. The microparticles can be degraded over time, inducing both secretory and systemic immune responses.

DETAILED DESCRIPTION:
Vaccine formulations of synthetic peptides adsorbed to alum may not provide other requisite characteristics of an effective HIV vaccine, such as induction of mucosal immunity, production of cytotoxic T cells, and ease of administration. An oral microparticulate vaccine containing a prototype synthetic peptide has been developed. The microparticles can be degraded over time, inducing both secretory and systemic immune responses.

Twelve volunteers per dose regimen will receive oral microparticulate multivalent HIV-1 peptide vaccine at months 0, 1, and 6, either daily as a low dose for 3 days or a single higher dose. Additionally, four volunteers per regimen will receive placebo. Volunteers are followed for 1 year. They will be contacted once or twice yearly for 5 years to check on health status.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* HIV negativity by ELISA within 8 weeks of study entry.
* Absolute CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.
* Lower or intermediate risk sexual behavior.

NOTE:

* No more than 10 percent of subjects may be over 50 years of age.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as psychosis or suicidal tendencies) or occupational responsibilities that preclude study compliance.
* Active syphilis. NOTE: Subjects whose serology is documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of anaphylaxis or other serious reactions to vaccines.
* History of inflammatory gastrointestinal disease, celiac disease, or intestinal malignancy.
* History of acute gastroenteritis within the past month or gastrointestinal surgery within the past year.
* History of cancer unless there has been surgical excision with reasonable assurance of cure.
* History of serious allergic reaction.

Prior Medication:

Excluded:

* History of immunosuppressive medications.
* Live attenuated vaccines within 60 days prior to study entry (NOTE: Medically indicated subunit or killed vaccines, e.g., influenza or pneumococcal, are not exclusionary, but should not be given within 2 weeks of HIV immunization).
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Identifiable higher risk behavior for HIV infection, including the following:

* History of injection drug use within the past 12 months.
* Higher risk sexual behavior as defined by the AVEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Overall Officials: Lambert J, Study Chair
Locations (2):
- United States (2):
  - Johns Hopkins Univ / Ctr for Immunological Research, Baltimore, Maryland
  - Univ of Rochester Med Ctr, Rochester, New York

REFERENCES:
- [Background] Kelleher AD, Emery S, Cunningham P, Duncombe C, Carr A, Golding H, Forde S, Hudson J, Roggensack M, Forrest BD, Cooper DA. Safety and immunogenicity of UBI HIV-1MN octameric V3 peptide vaccine administered by subcutaneous injection. AIDS Res Hum Retroviruses. 1997 Jan 1;13(1):29-32. doi: 10.1089/aid.1997.13.29. PMID 8989424
- [Background] Kahn J, Murcar N, Elbeik T, Staprans S, Hanson C, Mayer Y, Doyle R, Gonzalez L, Koff W. UBI HIV-1MN octameric V3 peptide vaccine in HIV-1 negative humans. Conf Adv AIDS Vaccine Dev. 1996 Feb 11-15:167 [Poster 47]